CLINICAL TRIAL: NCT00934245
Title: Direct and Indirect Protection by Influenza Vaccine Given to Children in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wayne Sullender, M.D. (Other)
Collaborators: All India Institute of Medical Sciences (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Wayne Sullender, M.D., Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F090422004; U01/IP000117-02
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: Influenza; India; Children; Trivalent Influenza Vaccine (TIV); Inactivated poliovirus vaccine (IPV); Direct vaccine effectiveness; Indirect vaccine effectiveness
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip; Poliovirus Vaccine, Inactivated; Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Inactivated Polio Vaccine (IPV) (Active Comparator): Inactivated trivalent poliovirus vaccine (IPV) age Dose # doses/year 1 # doses year 2 and 3 6 mo -8y 0.5 ml 2 1 9-10 y 0.5 ml 1 1
  Interventions: Biological: Inactivated polio vaccine (IPV)
- Inactivated Trivalent Influenza Vaccine (Experimental): Inactivated split virion trivalent influenza vaccine (TIV) age Dose # doses year 1 # doses year 2 and 3 6-35 mo 0.25 ml 2 1 3-8 y 0.5 ml 2 1 9-10 y 0.5 ml 1 1
  Interventions: Biological: Inactivated Trivalent Influenza Vaccine
- Surveillance arm (No Intervention): Those ineligible for vaccination will be enrolled for febrile acute respiratory illness (FARI) surveillance to assess indirect effects of vaccination in household members.

INTERVENTIONS:
Biological: Inactivated Trivalent Influenza Vaccine — Vaccine administration will occur twice, one month apart, in the first year of participation in the study. This will occur as TIV vaccine becomes available in India, in the early autumn. Subsequent years will provide one immunization. Due to the inclusion of the pandemic 2009 influenza A H1N1 virus in the 2010-2011 northern hemisphere vaccine formulation and recommendations that children should receive 2 doses of this vaccine this study will administer 2 doses of vaccine in the second year of the study.
  Other Names: split virion trivalent influenza vaccine, Vaxigrip
  Arms: Inactivated Trivalent Influenza Vaccine
Biological: Inactivated polio vaccine (IPV) — Vaccine administration will occur twice, one month apart, in the first year of participation in the study to parallel administration of TIV (experimental intervention). Subsequent years will provide one immunization except 2011 schedule modified to accommodate changes in TIV schedule as per above..
  Other Names: Imovax
  Arms: Inactivated Polio Vaccine (IPV)

SUMMARY:
The study described here will immunize children with trivalent influenza vaccine (TIV) and determine whether this reduces influenza illness among the immunized children and their older family members. The comparison or control group for the children receiving influenza vaccine will be children immunized with inactivated poliovirus vaccine (IPV). The study will also provide information on the amount of disease produced by influenza in the study population.

DETAILED DESCRIPTION:
Influenza is an important cause of illness among children and adults in the United States. Influenza is likely also an important cause of illness in India, but published data on influenza infections in India are limited, especially for children. Although influenza vaccines are used routinely in the United States, including in young children, influenza vaccines have not seen widespread use in India. This is likely due to the lack of information from India about disease burden due to influenza and because the influenza vaccines have never been tested for efficacy in India. In addition, because young children are thought to be important in the spread of influenza in families, it is possible immunization of children against influenza will reduce influenza infections among older children and adults in the home.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in either vaccine group (TIV or IPV) will require ages 6 months through 10 years of age.
* All individuals in enrolled households will be eligible for enrollment into surveillance arm.

Exclusion Criteria:

* Exclusion criteria from the vaccine groups includes known allergy to eggs, or hypersensitivity to other components of a vaccine (streptomycin, neomycin, and polymyxin B)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4598 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza infection in vaccinated child | 1 year

SECONDARY OUTCOMES:
Laboratory-confirmed influenza infection in household member of a vaccinated child | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Sullender, MD, Principal Investigator — University of Alabama at Birmingham; Shobha Broor, MD, Principal Investigator — All India Institute of Medical Sciences; Anand Krishnan, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Comprehensive Rural Health Services Project (CRHSP), Ballabgarh, Haryana, India

REFERENCES:
- [Background] Sullender W, Fowler K, Krishnan A, Gupta V, Moulton LH, Lafond K, Widdowson MA, Lal RB, Broor S. Design and initiation of a study to assess the direct and indirect effects of influenza vaccine given to children in rural India. Vaccine. 2012 Jul 27;30(35):5235-9. doi: 10.1016/j.vaccine.2012.06.002. Epub 2012 Jun 16. PMID 22709952
- [Background] Mir MA, Lal RB, Sullender W, Singh Y, Garten R, Krishnan A, Broor S. Genetic diversity of HA1 domain of hemagglutinin gene of pandemic influenza H1N1pdm09 viruses in New Delhi, India. J Med Virol. 2012 Mar;84(3):386-93. doi: 10.1002/jmv.23205. PMID 22246823
- [Derived] Sullender WM, Fowler KB, Gupta V, Krishnan A, Ram Purakayastha D, Srungaram Vln R, Lafond KE, Saha S, Palomeque FS, Gargiullo P, Jain S, Lal R, Widdowson MA, Broor S. Efficacy of inactivated trivalent influenza vaccine in rural India: a 3-year cluster-randomised controlled trial. Lancet Glob Health. 2019 Jul;7(7):e940-e950. doi: 10.1016/S2214-109X(19)30079-8. PMID 31200893